CLINICAL TRIAL: NCT00463411
Title: Study on Male Osteoporosis and Aging
Brief Title: Study of Male Osteoporosis and Aging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry); AP Moeller Foundation (Other)
Other Study IDs: 025
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2006-12

CONDITIONS: Osteoporosis
Keywords: osteoporosis; male; fracture risk; genetical epidemiology
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
The aim of this study is to identify potential risk factors for fragility fractures in men.

DETAILED DESCRIPTION:
Osteoporosis is a disease characterized by decreased bone mass and pathological changes in the microarchitecture of the bones. The clinical significance of osteoporosis is the association with fragility fractures and, consequently, increases in both morbidity and mortality.

In men, genetical and life-style factors are known to affect the risk of fractures, however, data relating these factors with measures of bone mineral density and fracture risk are limited.

30.000 men aged 60-70 were randomly selected from the Central Office of Civil Registration in Denmark. Each receive a questionnaire addressing demographics, potential risk factors of osteoporosis, past medical history and medication by mail. In case of consent, the participants will complete a full medical examination including DXA and sampling of DNA if they have a fragility fracture. At the same time, 2 participants from the study population will be selected as control. The study period is 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 60-70 being able to consent in writing

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30000
Dates: Start 2006-12; Study Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kim T Brixen, MD. Ph.d, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense, Denmark